CLINICAL TRIAL: NCT02649166
Title: Closing the Loop on Tremor: A Responsive Deep Brain Stimulator for the Treatment of Essential Tremor
Brief Title: Responsive Deep Brain Stimulator for Essential Tremor
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Medtronic (Industry); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201501021 -N-A; 5UH3NS095553-04 (NIH)
Record Dates: First submitted 2016-01-06; First posted 2016-01-07 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Essential Tremor
Keywords: Essential tremor; Kinetic tremor; Intention tremor
MeSH Terms: conditions — Essential Tremor; Tremor | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Deep brain stimulation (Experimental): All participants will undergo unilateral deep brain stimulation (DBS) implantation for essential tremor. Medtronic Summit RC+S devices will be used because these are capable of recording brain signals, as well as delivering DBS. Participants will receive continuous (open-loop) and closed-loop deep brain stimulation interventions, which will be compared for efficacy.
  Interventions: Device: Deep brain stimulation; Device: Closed-loop deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — The deep brain stimulation system includes an implantable neurostimulator, thalamic leads to be implanted in the ventral intermediate nucleus (Vim), and subdural cortical strips. The deep brain stimulation system will be set to provide continuous stimulation for the 6 months following surgery. Subjects will be seen monthly for evaluation as a part of normal clinical care for deep brain stimulation. At 6 months, the investigators will determine whether or not the subject is a candidate for closed-loop deep brain stimulation. Qualifying subjects will have the option to have their settings changed in order to participate in the RBS stimulation intervention. These subjects will been seen every 6 months for evaluation as part of normal clinical care for deep brain stimulation.
  Other Names: Medtronic Summit RC+S
Device: Closed-loop deep brain stimulation — The deep brain stimulation system includes an implantable neurostimulator, Vim thalamic leads, and subdural strips. Six months post-surgery, the deep brain stimulation system will be set to provide responsive stimulation for the duration of the study. Subjects will be seen every 6 months for evaluation as a part of normal clinical care for deep brain stimulation. Data gathered from the subject during the first 6 months will be used to determine if this intervention is applicable for each individual subject. Subjects who do not qualify will continue to receive the other study intervention.
  Other Names: Medtronic Nexus-E

SUMMARY:
Essential tremor is an incurable, degenerative brain disorder that results in increasingly debilitating tremor, and afflicts an estimated 7 million people in the US. In one study, 25% of essential tremor patients were forced to change jobs or take early retirement because of tremor. Essential tremor is directly linked to progressive functional impairment, social embarrassment, and even depression. The tremor associated with essential tremor is typically slow, involves the hands (and sometimes the head and voice), worsens with intentional movements, and is insidiously progressive over many years. Deep brain stimulation has emerged as a highly effective treatment for intractable, debilitating essential tremor. However, since the intention tremor of essential tremor is typically intermittent, and commonly absent at rest, the currently available continuous deep brain stimulation may be delivering unnecessary current to the brain that increases undesirable side effects such as slurred speech and walking difficulty, and hastens the depletion of device batteries, necessitating more frequent surgical procedures to replace spent pulse generators. The overall objective of this early feasibility study is to provide preliminary data on the safety and efficacy of "closed-loop" deep brain stimulation for intention tremor using novel deep brain stimulation devices capable of continuously sensing brain activity and delivering therapeutic stimulation only when necessary to suppress tremor.

DETAILED DESCRIPTION:
The purpose of this study is to investigate brain signals related to intention tremor in essential tremor in order to deliver deep brain stimulation only when the patient is showing symptoms. By delivering stimulation only when needed, the investigators hypothesize that the treatment will be more effective, will cause fewer adverse side effects and will increase battery time of the device (reducing the number of battery replacement surgeries).

Participation in this study will require extensive pre-surgical screening to determine eligibility for deep brain stimulation surgery, a deep brain stimulation surgical procedure, and regular follow-ups. Subjects will be seen monthly post surgery for 6 months. After 6 months, data will be assessed and closed-loop deep brain stimulation may be offered as a stimulation setting. If so, the stimulator settings will be changed from chronic to responsive. If not, the subject will continue to receive chronic deep brain stimulation stimulation. Subsequent visits will be scheduled every 6 months until a total of 24 months of study participation (also at month 9).

At the end of the initial 24-month study period, subjects will have the choice of 1) continuing active stimulation at the current setting, 2) continuing stimulation but searching for a new setting, 3) discontinuing stimulation (turning the device off), 4) having the device removed. If the subject continues to receive active stimulation, they will be followed by the investigators and seen at yearly intervals.

ELIGIBILITY:
Inclusion Criteria:

1. You provide informed consent.
2. You are over 21 years of age.
3. You are diagnosed with a postural-intention (essential) tremor for at least 3 years and meet strict diagnostic criteria and have been seen and examined by a movement disorders fellowship trained neurologist.
4. You have had a significant disabling medical-refractory upper extremity tremor with no evidence of supraspinal central nervous system disease or injury (tremor not adequately controlled by medications for at least three (3) months before implant).
5. You have had a postural or kinetic tremor severity score of at least 2 out of 4 in the extremity intended for treatment on the Fahn-Tolosa-Marin Clinical Rating Scale for Tremor (CRST).
6. You have had a CRST score of 2 or above in any one of the items 16-23 from the Disability subsection of the CRST: speaking, feeding other than liquids, bringing liquids to mouth, hygiene, dressing, writing, working and social activities.
7. Your tremor is refractory adequate trials of at least two medications, one of which should be either propranolol or primidone. An adequate medication trial is defined as a therapeutic dose of each medication or the development of side effects as the medication dose is titrated.
8. You are available for appropriate follow-up times for the length of the study.

Exclusion Criteria:

1. Any previous neurosurgical intervention including deep brain stimulation or ablative brain lesions.
2. Medication related movement disorders.
3. Any suspicion of Parkinsonian tremor, including presence of Parkinsonian features such as bradykinesia, rigidity, or postural instability.
4. Any behaviors consistent with ethanol or substance abuse as defined by the criteria outlined in DSM-V.
5. Severe medical co-morbidity including cardiovascular disorder, lung disorder, kidney disease, continuous neurological disease, hematological disease, or frailty that impact tolerability of the surgery as judged by the screening physicians.
6. Abnormal brain MRI including hydrocephalus, stroke, structural lesions, demyelinating lesions, or infectious lesions. Also excluded will be subjects with severe atrophy.
7. Any uncontrolled symptoms or signs of increased intracranial pressure (e.g., headache, nausea, vomiting, lethargy, papilledema).
8. A history of seizures within the past year.
9. A dementia rating scale score (DRS) <130 signifying significant cognitive dysfunction and a potential for inability to cooperate with tasks involved in the study.
10. Any attempt or intent of suicide in the last six months.
11. Presence or history of psychosis.
12. Significant or active mood disorders including depression. For the purpose of this study, we consider a significant mood disorder to include any subject who has:

    1. Scores ≥ 20 on the Patient Health Questionnaire - 9 (PHQ-9).
    2. Currently under the care of a psychiatrist
    3. Currently participating in cognitive-behavioral therapy
    4. Been hospitalized for the treatment of a psychiatric illness within 12 months
    5. Ever received transcranial magnetic stimulation
    6. Ever received electroconvulsive therapy

n. In addition, patients who are pregnant or plan to become pregnant will be excluded from this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Rating Scale for Tremor (CRST) for continuous deep brain stimulation | 6 months post-surgery
  - Reduction in Clinical Rating Scale for Tremor after 6 months as an effect of continuous Vim deep brain stimulation
  The Fahn-Tolosa-Marin Tremor Rating Scale is a clinical rating scale assessing severity of tremor by body part from 0 (none) to 4 (severe). The scale is divided into three parts, where Part A assesses tremor severity at rest, during posture, and kinetic maneuvers for nine body parts; Part B assesses ability to perform specific motor tasks/functions (writing, drawing, and pouring with dominant and nondominant hands); and Part C assesses patient-reported functional disability resulting from the tremor. Score ranges from 0 to 80 for Part A, from 0 to 36 for Part B, and from 0 to 28 for Part C. The total score obtained by adding the three parts is 144. A higher score indicates a higher severity of the tremor. Finally, the scale includes one separate item dealing with global assessment of tremor-related disability, rated by both patient and examiner on a 5-point scale.
Clinical Rating Scale for Tremor (CRST) for closed-loop deep brain stimulation | Baseline until 24 months post-surgery
  - Closed-loop deep brain stimulation as an effective alternative to continuous deep brain stimulation
  Clinical scores during continuous stimulation will be compared to scores on the during closed-loop stimulation.
Clinical Rating Scale for Tremor (CRST) for continuous deep brain stimulation | 24 months post-surgery
  - Reduction in Clinical Rating Scale for Tremor after 24 months as an effect of continuous Vim deep brain stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Gunduz, Ph.D, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Once 24 month follow-up is completed for all subjects, the investigators will consider data sharing requests for de-identified data.